CLINICAL TRIAL: NCT00016211
Title: Prophylactic Cranial Irradiation In Extensive Disease Small Cell Lung Cancer
Brief Title: Radiation Therapy to Prevent Brain Metastases in Patients With Previously Treated Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-22993-08993; EORTC-RA-22993; EORTC-LCG-08993
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Radiotherapy

INTERVENTIONS:
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Radiation therapy to the brain may be effective in preventing brain metastases. It is not yet known if radiation therapy is effective following chemotherapy in preventing brain metastases.

PURPOSE: Randomized phase III trial to determine the effectiveness of radiation therapy in preventing brain metastases in patients who have received chemotherapy for extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the incidence of, and time to, symptomatic brain metastases in patients with previously treated extensive stage small cell lung cancer treated with prophylactic cranial irradiation vs no further therapy.
* Compare the quality of life and survival of these patients.
* Determine the toxicity of this regimen in these patients.
* Determine the health economics associated with this study.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center and performance status. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Within 5 weeks after completion of prior chemotherapy, patients undergo prophylactic cranial irradiation once daily for 5-12 days.
* Arm II: Patients receive no further therapy after completion of prior chemotherapy.

Quality of life is assessed at baseline, 6 weeks, every 3 months for 1 year, and then every 6 months thereafter.

Patients are followed at 6 weeks, every 3 months for 1 year, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 287 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytologically or histologically confirmed small cell lung cancer

  * Documented extensive disease before the initiation of chemotherapy
* Responsive disease after 4 to 6 courses of initial chemotherapy

  * No more than 5 weeks since completion of prior chemotherapy
* No brain or leptomeningeal metastases

PATIENT CHARACTERISTICS:

Age:

* 18 to 75

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No other prior or concurrent malignancy except skin cancer or carcinoma in situ of the cervix
* No psychological, familial, sociological, or geographical condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics

Endocrine therapy:

* No concurrent corticosteroids

Radiotherapy:

* No prior radiotherapy to the brain
* No prior radiotherapy to the head and neck

Surgery:

* Not specified

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2001-02; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Time to symptomatic brain metastases measured by Logrank at 6 weeks, every 3 months in year 1, and then every 6 months

SECONDARY OUTCOMES:
Quality of life assessed by EORTC QLQ-C30 and EORTC BN-20 at baseline, 6 weeks, every 3 months in year 1, and then every 6 months
Toxicity assessed by NCI CTC v2.0 during treatment, at 6 weeks, every 3 months in year 1, and then every 6 months
Survival measured by Logrank at 6 weeks, every 3 months in year 1, and then every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: B.J. Slotman, PhD, MD, Study Chair — Free University Medical Center; Pieter E. Postmus, MD, Study Chair — Free University Medical Center
Locations (49):
- Belgium (6):
  - Ziekenhuis Netwerk Antwerpen Middelheim, Antwerp
  - Universiteit Gent, Ghent
  - Hopital de Jolimont, Haine-Saint-Paul
  - Cazk Groeninghe - Campus Maria's Voorzienigheid, Kortrijk
  - Centre Hospitalier Regional de la Citadelle, Liège
  - Clinique Saint-Joseph, Liège
- Bank Of Cyprus Oncology Centre, Nicosia, Cyprus
- National Cancer Institute of Egypt, Cairo, Egypt
- Institut Gustave Roussy, Villejuif, France
- Universitaetsklinikum Hamburg-Eppendorf, Hamburg, Germany
- University of Kaposvar, Kaposvár, Hungary
- Rambam Medical Center, Haifa, Israel
- Italy (3):
  - Ospedale Santa Croce, Cuneo
  - Istituto Nazionale per la Ricerca sul Cancro, Genoa (Genova)
  - Azienda Ospedaliera Di Parma, Parma
- Netherlands (11):
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Academisch Medisch Centrum at University of Amsterdam, Amsterdam
  - Arnhems Radiotherapeutisch Instituut, Arnhem
  - Radiotherapeutisch Instituut-(Riso), Deventer
  - University Medical Center Groningen, Groningen
  - Radiotherapeutisch Instituut Friesland, Leeuwarden
  - Leiden University Medical Center, Leiden
  - Nijmegen Cancer Center at Radboud University Medical Center, Nijmegen
  - University Medical Center Rotterdam at Erasmus Medical Center, Rotterdam
  - Erasmus MC - Sophia Children's Hospital, Rotterdam
  - Dr. Bernard Verbeeten Instituut, Tilburg
- Medical University of Gdansk, Gdansk, Poland
- Marmara University Hospital, Istanbul, Turkey (Türkiye)
- United Kingdom (21):
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Princess Royal Hospital, Hull, England
  - Cookridge Hospital at Leeds Teaching Hospital NHS Trust, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Christie Hospital N.H.S. Trust, Manchester, England
  - Clatterbridge Centre for Oncology NHS Trust, Merseyside, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Royal Shrewsbury Hospital, Shrewsbury, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Southend NHS Trust Hospital, Westcliff-on-Sea, England
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Western Infirmary, Glasgow, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Nevill Hall Hospital, Gwent, Wales
  - Royal Gwent Hospital, Newport Gwent, Wales

REFERENCES:
- [Result] Slotman BJ, Mauer ME, Bottomley A, Faivre-Finn C, Kramer GW, Rankin EM, Snee M, Hatton M, Postmus PE, Collette L, Senan S. Prophylactic cranial irradiation in extensive disease small-cell lung cancer: short-term health-related quality of life and patient reported symptoms: results of an international Phase III randomized controlled trial by the EORTC Radiation Oncology and Lung Cancer Groups. J Clin Oncol. 2009 Jan 1;27(1):78-84. doi: 10.1200/JCO.2008.17.0746. Epub 2008 Dec 1. PMID 19047288
- [Result] Slotman B, Faivre-Finn C, Kramer G, et al.: A randomized trial of prophylactic cranial irradiation (PCI) versus no PCI in extensive disease small cell lung cancer after a response to chemotherapy (EORTC 08993-22993). [Abstract] J Clin Oncol 25 (Suppl 18): A-4, 2s, 2007.
- [Result] Slotman B, Faivre-Finn C, Kramer G, Rankin E, Snee M, Hatton M, Postmus P, Collette L, Musat E, Senan S; EORTC Radiation Oncology Group and Lung Cancer Group. Prophylactic cranial irradiation in extensive small-cell lung cancer. N Engl J Med. 2007 Aug 16;357(7):664-72. doi: 10.1056/NEJMoa071780. PMID 17699816
- [Result] Slotman BJ, Faivre-Finn C, Kramer GWPM, et al.: Prophylactic cranial irradiation (PCI) in extensive stage small cell lung cancer (ES-SCLC) (EORTC 22993-08993). [Abstract] Int J Radiat Oncol Biol Phys 69 (3 Suppl): A-7, S4, 2007.
- [Derived] Bernhardt D, Adeberg S, Bozorgmehr F, Opfermann N, Hoerner-Rieber J, Repka MC, Kappes J, Thomas M, Bischoff H, Herth F, Heussel CP, Debus J, Steins M, Rieken S. Nine-year Experience: Prophylactic Cranial Irradiation in Extensive Disease Small-cell Lung Cancer. Clin Lung Cancer. 2017 Jul;18(4):e267-e271. doi: 10.1016/j.cllc.2016.11.012. Epub 2016 Dec 2. PMID 28027850
- [Derived] Slotman BJ, Faivre-Finn C, Kramer GW, Rankin E, Snee M, Hatton M, Postmus PE, Collette L, Musat E, Senan S. [Prophylactic cranial irradiation in patients with extensive disease caused by small-cell lung cancer responsive to chemotherapy: fewer symptomatic brain metastases and improved survival]. Ned Tijdschr Geneeskd. 2008 Apr 26;152(17):1000-4. Dutch. PMID 18549175